CLINICAL TRIAL: NCT03209271
Title: Hemodynamic Effects of Cold Versus Warm Fluid Bolus Infusion in Healthy Volunteers: a Randomized Cross-over Trial
Brief Title: Hemodynamic Effects of Cold Versus Warm Fluid Bolus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Christer Svensen, Professor, Karolinska Institutet
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: EPN 2016/986-31/1
Record Dates: First submitted 2017-06-26; First posted 2017-07-06 (Actual); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Temperature Change, Body; Hypovolemia
Keywords: Fluid therapy
MeSH Terms: conditions — Body Temperature Changes; Hypovolemia | interventions — Ringer's acetate; Cold Temperature

STUDY DESIGN:
Intervention Model Description: Crossover study of 2 different temperatures of crystalloid fluid bolus.
Masking Description: Unblinded (unable to blind subjects)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Body temperature fluid (Experimental): 500ml Ringers Acetate infused over 15 minutes warmed to 38°C
  Interventions: Drug: Ringer's Acetate (warm)
- Room temperature fluid (Active Comparator): 500ml Ringers Acetate infused over 15 minutes cooled to 22°C
  Interventions: Drug: Ringer's Acetate (cold)

INTERVENTIONS:
Drug: Ringer's Acetate (warm) — Body temperature fluid
  Other Names: Ringer-Acetat Baxter Viaflo, ATC B05BB01
  Arms: Body temperature fluid
Drug: Ringer's Acetate (cold) — Room temperature fluid
  Other Names: Ringer-Acetat Baxter Viaflo, ATC B05BB01
  Arms: Room temperature fluid

SUMMARY:
Fluid boluses are often administered with the aim of improving tissue perfusion in critically ill patients. It is unclear whether the temperature of the fluid has an impact on the hemodynamic response. The aim of this study is to describe the hemodynamic effects of a fluid bolus with two different temperatures.

DETAILED DESCRIPTION:
A randomized, controlled, cross-over study in 21 healthy volunteers. The participants will receive a fluid bolus of 500 ml Ringer's Acetate at either 22°C or 38°C over 15 minutes in a randomized order. Non-invasive measures will be made of cardiac index, mean arterial pressure, systolic blood pressure, diastolic blood pressure, heart and pulse rate, saturation and temperature. Hemodynamic measure will be made using the Clearsight® system. Measurements will be made during 120 minutes. The second session will take place at least one day later, and the participant will then receive the other fluid temperature.

ELIGIBILITY:
Inclusion Criteria:

- Volunteers 18 years or older Previously healthy

Exclusion Criteria:

* American Society of Anesthesiologists classification 2 or above.
* Known pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-02-03 (Actual); Primary Completion 2017-05-27 (Actual); Study Completion 2017-05-27 (Actual)

PRIMARY OUTCOMES:
Cardiac index 15 minutes | 15 minutes
  Change in cardiac index at 15 minutes from start of infusion

SECONDARY OUTCOMES:
Cardiac index 120 minutes | 120 minutes
  Change in cardiac index during 120 minutes from start of infusion
Blood pressure 120 minutes | 120 minutes
  Change in blood pressure during 120 minutes from start of infusion
Heart rate 120 minutes | 120 minutes
  Change in heart rate during 120 minutes from start of infusion
Temperature 120 minutes | 120 minutes
  Change in body temperature during 120 minutes from start of infusion

OTHER OUTCOMES:
Time to return to baseline for CI | 0-120 minutes
  Time to return to baseline for CI
Time to return to baseline for blood pressure | 0-120 minutes
  Time to return to baseline for blood pressure
Time to return to baseline for heart rate | 0-120 minutes
  Time to return to baseline for heart rate
Time to return to baseline for temperature | 0-120 minutes
  Time to return to baseline for temperature

CONTACTS AND LOCATIONS:
Overall Officials: Maria Cronhjort, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet Södersjukhuset, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wall O, Ehrenberg L, Joelsson-Alm E, Martensson J, Bellomo R, Svensen C, Cronhjort M. Haemodynamic effects of cold versus warm fluid bolus in healthy volunteers: a randomised crossover trial. Crit Care Resusc. 2018 Dec;20(4):277-284. PMID 30482135